CLINICAL TRIAL: NCT03860545
Title: The New Biochemical Markers of Cardiac Surgery Related Acute Kidney Injury.
Brief Title: New Markers of Cardiac Surgery Related Acute Kidney Injury.
Status: Completed | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Jowita Biernawska, MD PhD, Pomeranian Medical University Szczecin
Other Study IDs: KB - 0012/146/10
Record Dates: First submitted 2019-02-26; First posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Acute Kidney Injury; Cardiac Disease
Keywords: Acute Kidney Injury, cardiopulmonary bypass; brush-border enzymes of the proximal renal tubules; ischemia modified albumin
MeSH Terms: conditions — Acute Kidney Injury; Heart Diseases | interventions — Urination; Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-AKI: patient without acute kidney injury (AKI) during perioperative observation period
  Interventions: Diagnostic Test: urine and blood analysis
- AKI: patient with diagnosis acute kidney injury (AKI) established during perioperative observation period
  Interventions: Diagnostic Test: urine and blood analysis

INTERVENTIONS:
Diagnostic Test: urine and blood analysis — concentration of ischemia modified albumin assessed in blood before operation, immediately and one hour after cardiopulmonary bypass, 24 hours after operation; concentration of urinary excretion of brush-border enzymes of the proximal renal tubules assessed before operation, immediately and one hour after cardiopulmonary bypass, 24 hours after operation, serum creatinine levels will be evaluated on the day of the operation and 24 h and 48 h postoperatively

SUMMARY:
Cardiac surgery related acute kidney injury (CS-AKI) is a clinical problem associated with a cardiopulmonary bypass used during cardiac surgery procedures. In this study the investigators will assess the biochemical markers of acute kidney injury such as ischemia modified albumin (IMA) or urinary excreted of brush-border enzymes of the proximal renal tubules perioperatively. There has been no official recommendations toward routine use of analysed biomarkers.

DETAILED DESCRIPTION:
Cardiac surgery related acute kidney injury (CS-AKI) is an important clinical problem. Kidney injury occurs following a cardiopulmonary bypass used during cardiac surgery procedures. The pathomechanisms of acute kidney injury (AKI) is complex and multifactorial. It may involve few injury pathways: ischemia and reperfusion, endogenous toxins, inflammation, metabolic factors and oxidative stress. Biochemical markers of acute kidney injury such as ischemia modified albumin (IMA) or urinary excreted of brush-border enzymes of the proximal renal tubules analysed perioperatively will be assessed in this study. There has been no official recommendations toward routine use of analysed biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* a planned operation of coronary artery bypass grafting with the use of cardiopulmonary bypass

Exclusion Criteria:

* emergency operations or re-operations;
* a known pathology of the urinary tract or renal failure;
* chronic use of the following medications: iron, non-steroidal anti-inflammatory drugs (NSAIDs), immunosuppression, or steroids in the preoperative period;
* polycythemia, porphyria or pathological hemoglobin species in anamnesis;
* preoperative signs of hepatic failure;
* active autoimmune or neoplastic diseases, active infection;
* anticipated significant bleeding (anti-platelet agents), suggesting the use of blood-derived products during the operation and afterward
* acute myocardial infarction after operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be divided into 2 groups regarding postoperative acute kidney injury
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
acute kidney injure after operation | up to 48 hours post operation
  acute kidney injure measured by creatinine concentration mg/dl
acute kidney injure after operation | up to 48 hours post operation
  acute kidney injure measured by urine output in ml

CONTACTS AND LOCATIONS:
Locations (1):
- Pomeranian Medical University, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: Undecided
encoded in database of principal investigator